CLINICAL TRIAL: NCT03314714
Title: The Dual Role of Intramyocellular Lipids in Mediating Insulin Resistance: Assessing the Mechanisms of the Athlete's Paradox
Brief Title: Duality of Lipids: the Athlete's Paradox
Acronym: LIDDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Diabetes Center (Other)
Collaborators: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DDZ-LIDDIA01
Record Dates: First submitted 2017-04-03; First posted 2017-10-19 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Insulin Resistance, Diabetes; Lipid Metabolism Disorders
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus; Lipid Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute bout of endurance exercise (Experimental): Intramyocellular lipid metabolism will be assessed in insulin resistant and healthy, sedentary individuals after an acute bout of endurance exercise.
  Interventions: Procedure: Acute bout of endurance exercise

INTERVENTIONS:
Procedure: Acute bout of endurance exercise — Individuals will undergo an acute bout of endurance exercise for 90 min at 75% of maximal oxygen uptake.

SUMMARY:
Accumulation of intramyocellular lipids (IMCLs) due to increased supply of fatty acids can induce defects in the insulin signaling cascade, causing skeletal muscle insulin resistance. However, the causes for muscle insulin resistance are not well understood. The association of elevated IMCLs and insulin resistance has been shown in obese humans and individuals with type 2 diabetes as well as several animal models of insulin resistance. Despite the strong relationship between IMCLs and insulin resistance, this suggested relationship disappears when well-trained endurance athletes are included into this consideration as this group is highly insulin sensitive. This metabolic enigma has been termed the 'athlete's paradox'. The aim of this project is to resolve the mechanisms contributing to the athlete's paradox.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is characterized by an increasing insensitivity of muscle, fat and liver cells to the hormone insulin. About 9% of the global population is affected by this condition and mortality risk is twice as high in individuals with diabetes compared to similar-aged people without diabetes.

Muscle is of particular importance for glucose homeostasis, since in healthy subjects it accounts for 80-90% of postprandial insulin-stimulated glucose disposal. After cellular uptake of glucose by the specialized glucose transporter 4 (GLUT4), glucose is phosphorylated and stored as glycogen. In individuals with obesity or T2D, the capacity for insulin to facilitate glucose uptake and glycogen synthesis is impaired. This reduced response of a given insulin concentration to exert its biological effect is termed insulin resistance. Subsequent diminished insulin secretion due to β-cell failure results in fasting hyperglycemia and overt diabetes. Importantly, muscle insulin resistance is the initial defect occurring in the development of T2D and precedes the clinical development of the disease by up to 20 years. Intracellular defects in glucose transport have been identified as the limiting step for insulin-mediated glucose uptake into skeletal muscle. Impaired muscle glucose transport activity is likely a consequence of ectopic lipid accumulation and subsequent dysregulation of intramyocellular fatty acid metabolism. Indeed, results from normal weight, nondiabetic adults suggest that intramyocellular triglyceride content is a strong predictor for muscle insulin resistance. Of note, the development of insulin resistance occurred without changes in intramyocellular triglyceride content, thus dissociating the amount of these neutral storage lipids from insulin resistance. Instead, the bioactive lipid species diacylglycerols (DAG) and ceramides have been implicated in interfering with insulin signaling and glucose homeostasis in obese and insulin resistant individuals and individuals with T2D by activating members of the protein kinase C (PKC) family while ceramides mediate an increase in protein phosphatase 2A (PP2A) and an association of PKCζ and protein kinase B (PKB)/Akt2. To add another layer of complexity, DAGs seem to exert their detrimental intracellular effects in a subspecies- (mostly C18:0, C18:1, or C18:2 DAGs) and stereo-selective manner (sn-1,2 stereoisomer DAG). Taken together, excessive amounts of bioactive intramyocellular lipids (IMCLs) contribute to defective insulin signaling in obese individuals and patients with T2D. Surprisingly, endurance athletes have comparable amounts of IMCLs, but remain highly insulin sensitive. This metabolic conundrum has been termed "athlete's paradox".

This study therefore aims at resolving this conundrum with mass-spectrometry based state-of-the-art methodology by analysing lipid subspecies in endurance-trained athletes, untrained healthy individuals and insulin-resistant individuals.

ELIGIBILITY:
Inclusion criteria

* Insulin-resistant, non-athletic persons with a comparable content of IMCLs as the athletes
* Healthy, insulin-sensitive, normal-weight, non-athletic (BMI 18-25 kg / m2) individuals
* Endurance trained individuals (VO2max≥60 mL / kg / min ♂ and 45 mL / kg / min ♀)
* Male and female, age between ≥ 18 and ≤ 69 years

Exclusion criteria

* Acute infections / fever
* Immunosuppressive therapy
* Serious heart, kidney or liver disease: - New York Heart Association-Classification (NYHA) stage ≥ II - creatinine ≥ 1.6 mg / dl - Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≥ two-fold upper reference value - severe peripheral artery disease (PAD) (stage IV)
* autoimmune diseases
* Anemia (Hb <12g / l)
* Severe psychiatric illness or addiction
* Malignant cancer
* Participation in another intervention study
* Blood clotting disorders or increased risk of thrombosis
* Pregnancy, lactation
* Cigarettes (or non-smokers <1 year)
* alcohol consumption (men> 30g / d, women> 20g / d)
* ECG changes (ST reductions or - elevations, high-grade rhythm disorders (salvage or polytope extrasystoles, ventricular tachycardia)
* Heart diseases (angina pectoris at rest or under light load, myocardial infarction, thromboembolic processes / pulmonary embolism or severe arteriosclerosis, acute myocarditis or pericarditis, cardiac wall aneurysms, cor pulmonale, aortic stenosis)
* Hypertension (> 220/120 mmHg)
* Pacemaker
* Metallic and magnetic implants (for example, mechanical heart valves, joint prostheses, clip after vascular surgery, middle and inner ear implants or fresh dental implants, penis implants)
* Waist circumference> 135cm
* Claustrophobia

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Assessment of intramyocellular lipid content via magnetic resonance spectroscopy | 2 years
  Intramyocellular lipid content assessed via magnetic resonance spectroscopy (%lipid) in endurance-trained athletes and sedentary individuals
Assessment of intramyocellular lipid composition via mass spectrometry | 2 years
  Detailed composition of intramyocellular lipids assessed via mass spectrometry (concentration of bioactive lipids) in endurance-trained athletes and sedentary individuals

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof., MD, Principal Investigator — German Diabetes Center
Locations (2):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goodpaster BH, He J, Watkins S, Kelley DE. Skeletal muscle lipid content and insulin resistance: evidence for a paradox in endurance-trained athletes. J Clin Endocrinol Metab. 2001 Dec;86(12):5755-61. doi: 10.1210/jcem.86.12.8075. PMID 11739435
- [Background] Roden M, Price TB, Perseghin G, Petersen KF, Rothman DL, Cline GW, Shulman GI. Mechanism of free fatty acid-induced insulin resistance in humans. J Clin Invest. 1996 Jun 15;97(12):2859-65. doi: 10.1172/JCI118742. PMID 8675698
- [Background] Szendroedi J, Yoshimura T, Phielix E, Koliaki C, Marcucci M, Zhang D, Jelenik T, Muller J, Herder C, Nowotny P, Shulman GI, Roden M. Role of diacylglycerol activation of PKCtheta in lipid-induced muscle insulin resistance in humans. Proc Natl Acad Sci U S A. 2014 Jul 1;111(26):9597-602. doi: 10.1073/pnas.1409229111. Epub 2014 Jun 16. PMID 24979806
- [Derived] Pesta D, Anadol-Schmitz E, Sarabhai T, Op den Kamp Y, Gancheva S, Trinks N, Zaharia OP, Mastrototaro L, Lyu K, Habets I, Op den Kamp-Bruls YMH, Dewidar B, Weiss J, Schrauwen-Hinderling V, Zhang D, Gaspar RC, Strassburger K, Kupriyanova Y, Al-Hasani H, Szendroedi J, Schrauwen P, Phielix E, Shulman GI, Roden M. Determinants of increased muscle insulin sensitivity of exercise-trained versus sedentary normal weight and overweight individuals. Sci Adv. 2025 Jan 3;11(1):eadr8849. doi: 10.1126/sciadv.adr8849. Epub 2025 Jan 1. PMID 39742483